CLINICAL TRIAL: NCT07147790
Title: Comparative Study of Negative-Pressure Wound Therapy Integrated With Silver Nanoparticle Spray Versus Negative-Pressure Wound Therapy in Post-Revascularization Diabetic Foot Wound Management
Acronym: SNIPS-FOOT
Status: Enrolling by invitation | Type: Observational
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohab Mohamed Abdelfattah Saeed, Lecturer, Kafrelsheikh University
Other Study IDs: KFSIRB200-252; medical_research@kfs.edu.eg (Other: kafrelsheikh university)
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Ischemia Limb; Diabete Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- two groups A and B groups: A total of 100 patients were randomized into two equal groups using a computer-generated list with sealed opaque envelopes. Twelve patients were excluded post-randomization, resulting in 88 patients (44 per group) for final analysis.
  Group A received NPWT integrated with silver nanoparticle spray applied for 15 minutes before NPWT application using foam pre-soaked with the same spray. Group B received standard NPWT after saline irrigation. NPWT settings were -125 mmHg, continuous, with dressing changes every 72 hours.
  Interventions: Drug: After successful revacularization, We will categorize patients into two groups : groups A (The patient's wound will be cleaned and irrigated with silver nanoparticle spray, then we will cover the woun; Drug: Silver Nanoparticles Irrigant

INTERVENTIONS:
Drug: After successful revacularization, We will categorize patients into two groups : groups A (The patient's wound will be cleaned and irrigated with silver nanoparticle spray, then we will cover the woun — After successful revacularization, We will categorize patients into two groups :
  groups A (The patient's wound will be cleaned and irrigated with silver nanoparticle spray, then we will cover the wound with silver nanoparticle spray for 15 minutes (time needed for its absorption) before applying NPWT with foam soaked in silver nanoparticle spray) and group B (The patient's wounds will be cleaned and irrigated with a normal saline solution for 15 minutes before applying NPWT.). Standard NPWT setting will be used in both groups, with a continuous negative pressure range from 70 to 125 mmHg. Selection criteria for the application of VAC therapy will be presented by calcaneal, dorsal, or plantar foot ulcers with an area of 4.0 and 10.2 cm2. The NPWT dressing will be changed every 3 days. The endpoint of NPWT will be the appearance of healthy granulation tissue.
Drug: Silver Nanoparticles Irrigant — After successful revacularization, We will categorize patients into two groups :
  groups A (The patient's wound will be cleaned and irrigated with silver nanoparticle spray, then we will cover the wound with silver nanoparticle spray for 15 minutes (time needed for its absorption) before applying NPWT with foam soaked in silver nanoparticle spray) and group B (The patient's wounds will be cleaned and irrigated with a normal saline solution for 15 minutes before applying NPWT.). Standard NPWT setting will be used in both groups, with a continuous negative pressure range from 70 to 125 mmHg. Selection criteria for the application of VAC therapy will be presented by calcaneal, dorsal, or plantar foot ulcers with an area of 4.0 and 10.2 cm2. The NPWT dressing will be changed every 3 days. The endpoint of NPWT will be the appearance of healthy granulation tissue.

SUMMARY:
This was a prospective, parallel-group, randomized controlled trial conducted at the Vascular Surgery Department of Kafrelsheikh University Hospital, Egypt. The study was approved by the Institutional Review Board and conducted in accordance with the Declaration of Helsinki. Written informed consent was obtained from all participants.

Patients were eligible if they were ≥18 years of age, had diabetes mellitus with critical limb ischemia (CLI) classified as Rutherford category 6 or Fontaine stage IV, and presented with infected or ischemic foot wounds (Wagner grades 2-4) after successful revascularization confirmed by clinical and imaging evaluation. Exclusion criteria included osteomyelitis, active purulent discharge requiring further debridement, known allergy to silver or NPWT components, and inability to attend follow-up.

A total of 100 patients were randomized into two equal groups using a computer-generated list with sealed opaque envelopes. Twelve patients were excluded post-randomization, resulting in 88 patients (44 per group) for final analysis.

Group A received NPWT integrated with silver nanoparticle spray applied for 15 minutes before NPWT application using foam pre-soaked with the same spray. Group B received standard NPWT after saline irrigation. NPWT settings were -125 mmHg, continuous, with dressing changes every 72 hours.

Primary outcome: time to complete epithelialization. Secondary outcomes: wound size reduction, CRP change, infection rate, pain (VAS), hospital stay, reintervention.

Patients were followed weekly for 1 month and then biweekly for 6 months. CRP, WBC, wound measurements, and VAS were assessed at each visit.

SPSS v26 was used for analysis. Shapiro-Wilk test for normality. Independent t-tests and Mann-Whitney U tests for continuous data. Chi-square or Fisher's exact test for categorical variables. Significance at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patient with critical limb ischemia(CLI) Rutherford stage 6 or Fontaine stage 4. Wounds classified as Wagner classification grade 2 to 4.Successful revascularization was confirmed by imaging and clinical assessment.

Exclusion Criteria:

- 1. Patients with active infection(pus discharge and still need debridement), osteomyelitis.

2. patients who are allergic to silver or any components used in NPWT. 3. patients who are unable to follow up with us. patient

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients patient with peripheral arterial disease CLI RUTHERFORD 6,5
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
time to complete wound healingduring | during 1 year follow up period

CONTACTS AND LOCATIONS:
Locations (1):
- Kafr El Shaykh University, Kafr ash Shaykh, Kafrelshaykh Governorate, Egypt